CLINICAL TRIAL: NCT04136574
Title: Hand Dermatitis in the Care and Hospital Staff of the Brest CHRU: State of Play
Brief Title: Hand Dermatitis in the Care and Hospital Staff
Acronym: MANUS-PRO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0132
Record Dates: First submitted 2019-08-05; First posted 2019-10-23 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Hand Dermatoses
Keywords: hand dermatoses; hand dermatitis; occupationnal; caregivers; hand hygiene
MeSH Terms: conditions — Hand Dermatoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of the prevalence and risk factors of occupational dermatitis in the hands of caregivers and hospital staff of the Brest CHRU.

DETAILED DESCRIPTION:
Monocentric cross-sectional descriptive study by anonymous self-questionnaire designed to evaluate among caregivers and agents hospitals of the CHRU de Brest:

* the prevalence of occupational hands dermatitis
* the risk factors for hands dermatitis
* the clinical description of the hands dermatitis
* the rates of dermatitis according to hand hygiene practices (soap, hydro-alcoholic solution, associations of the two, wearing gloves ...)
* the changes in the hygiene practices of caregivers and hospital staff of the University Hospital caused by hand dermatitis.
* the professional and socio-economic impact of these hands dermatitis
* the evaluation of the use of care for these hands dermatitis.
* the assessment of the association of hand dermatitis with a personal or family atopic history.

ELIGIBILITY:
Inclusion Criteria:

* Any caregiver, hospital staff or staff involved incare or stretchering of CHU patients returning tosocioprofessional categories cited in the questionnaire.
* Major person
* Participation Agreement

Exclusion Criteria:

* Minor person.
* Administrative Services Staff, Restaurant Staff,technical staff
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Personal medical and paramedical caregivers and hospital staff working at the University Hospital ofBrest (any site confused). This population therefore includes: doctors, midwives,nurses or specialized nurses, caregivers, hospital service officers, studentshealth, dentists, physiotherapists and other paramedical professions.
Sampling Method: Non-Probability Sample
Enrollment: 1138 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
prevalence of occupational hands dermatitis | Three months (at the end of study)
  prevalence of occupational hands dermatitis among the staff of the Brest CHRU.

SECONDARY OUTCOMES:
Risk Factors for Hand Dermatitis | Three months (at the end of study)
  Risk Factors for Hand Dermatitis in Caregivers and Hospital Workers of the Brest Hospital
Clinical description of the dermatitis of the hands | Three months (at the end of study)
  Clinical description of the dermatitis of the hands of the caregivers and the hospital agents of the CHRU of Brest.
rate of dermatitis according to the hygiene practices | Three months (at the end of study)
  rate of dermatitis according to the hygiene practices of the hands (soap, SHA, combinations of both, wearing gloves ...)
changes in hygiene practices | Three months (at the end of study)
  changes in hygiene practices caregivers and hospital staff of the hospital induced by hands dermatitis
Assessment of the professional and socio-economic impact of hand dermatitis | Three months (at the end of study)
  Assessment of the professional and socio-economic impact of hand dermatitis in the care and hospital staff of the Hospital.
Assessment of the use of care for these hand dermatitis | Three months (at the end of study)
  Assessment of the use of care for these hand dermatitis
atopic status | Three months (at the end of study)
  atopic status
Percentage, means, and standard deviations of responses to quantitative and qualitative questions that appeal to the primary and secondary objectives. | Three months (at the end of study)
  Percentage, means, and standard deviations of responses to quantitative and

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France